CLINICAL TRIAL: NCT01048632
Title: A Pilot Study of the Safety and Efficacy of Oxandrolone in the Prevention and Treatment of Malnutrition in Infants After Cardiac Surgery
Brief Title: Pilot Study of the Safety and Efficacy of Oxandrolone in the Prevention and Treatment of Malnutrition in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Phillip Burch, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41510
Record Dates: First submitted 2010-01-08; First posted 2010-01-13 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition
Keywords: Neonates with HLHS or variant with plan to undergo Norwood Procedure
MeSH Terms: conditions — Malnutrition | interventions — Oxandrolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxandrolone (Experimental): Following clinical evaluation, all patients will be receive oxandrolone in addition to their usual medications. Based upon the patient's body weight, the coordinator, PI or sub-PI will determine the appropriate dose of oxandrolone (0.1 mg/kg/dose twice daily via the buccal mucosa.)
  Interventions: Drug: Oxandrolone

INTERVENTIONS:
Drug: Oxandrolone — 2.5 mg oxandrolone tablets.Based upon the patient's body weight, the coordinator, PI or sub-PI will determine the appropriate dose of oxandrolone (0.1 mg/kg/dose twice daily via the buccal mucosa.)

SUMMARY:
Oxandrolone is an anabolic steroid, marketed in the United States as an adjunctive therapy to combat weight loss resulting from chronic infection, extensive surgery, severe trauma, protein catabolism associated with prolonged administration of corticosteroids, and for the relief of bone pain accompanying osteoporosis. In children, it has been used to prevent and treat growth failure associated with severe burns (≥ 40% of total body surface area), Duchenne muscular dystrophy, Turner's syndrome, constitutional delay of growth and puberty, and chronic wasting in HIV-positive pediatric patients. Other applications in children have included treatment of central idiopathic precocious puberty, hereditary angioedema, and bilateral congenital anorchia. Growth failure is a common feature of infants with complex congenital heart disease, and can adversely affect outcome. This therapy has not been previously implemented in neonates thus we will evaluate the safety and efficacy of administering oxandrolone to improve growth in neonates with complex congenital heart disease who have undergone surgical palliation or repair by collecting anthropometric measurements and pharmacokinetic data.

Neonates with HLHS or variant with planned Norwood Procedure. The primary aims of this pilot study are to assess safety and efficacy of oxandrolone in this population. Our goal will be to enroll 5 patients in each phase of this pilot study. The incidence of adverse events will also be monitored and compared to untreated patients. Enrollment will continue until the target of 20 total patients has been met.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with HLHS, with plan to undergo the Norwood Procedures

Exclusion Criteria:

* Neonates with a birth weight ≤2.5 kg and gestational age ≥38 weeks (indicating intrauterine growth retardation), gestational age < 35 weeks (premature infants), and/or chromosomal or recognizable phenotypic syndrome of non-cardiac congenital abnormalities associated with growth failure (e.g. Trisomy 21, Trisomy 13, Noonan's syndrome, Turner's syndrome) will be excluded from enrollment. Neonates who will not be placed on the high risk feeding protocol postoperatively will also be excluded.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
PK testing | 48 hours

SECONDARY OUTCOMES:
Measures of Severity of Malnutrition to include pre albumin, C-reactive protein, nitrogen balance and measurements of somatic growth. | Measurements: Baseline, Day #1, Day #7, Day #14, Day #21, Day #28

CONTACTS AND LOCATIONS:
Overall Officials: Phillip T Burch, MD, Principal Investigator — University of Utah Dept. of Surgery-Div Cardiothoracic surgery
Locations (1):
- Primary Childrens Hospital, Salt Lake City, Utah, United States